CLINICAL TRIAL: NCT00958490
Title: Effects of a Physical Activity Intervention Walking Program on Quality of Life, Physical Activity Monitoring, and Functional Status of Post-Surgical Lumbar Spinal Stenosis Patients
Brief Title: Effects of a Walking Program on Functional Status of Post-Surgical Lumbar Spinal Stenosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Responsible Party: Dr. Michael Johnson/Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2006:040
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

ARMS (2):
- First walking group (Active Comparator): Group walking at 2 months postop
  Interventions: Other: Walking program
- Second group walking (Active Comparator): Group walking at 3 months postop
  Interventions: Other: Walking program

INTERVENTIONS:
Other: Walking program — 4 week physical activity walking program

SUMMARY:
Overall Objective: To evaluate the efficacy of an interventional walking program on the quality of life and functional status of patients with Lumbar Spinal Stenosis, post-surgery, using subjective (VAS, ODI, RMDQ, SF-36), and objective measures (triaxial accelerometry, step count, weight).

Design and Methods: Two groups of subjects will be examined; patients diagnosed with lumbar spinal stenosis (LSS) that progress to surgical management, with one group of subjects staring on the walking program at 2 months postop, and the other group starting on the walking program at 3 months postop.

Subjects who agree to participate will be assessed (assessments listed below) after the diagnosis preoperatively and 2 months postoperatively. One half of the group will start the walking program at the 2 months postop visit and be assessed again at the end of the walking program, the other half will be assessed again at 3 months postop and start the walking program at that time and be assessed again at 4 months postop. All subjects will be contacted by phone during their walking program to allow for questions from the subjects and to offer support and encouragement. Subjects will be given instructions and a daily diary to track steps taken each day (appendix A).

Subjects will be recruited from the referrals to the practices of the Orthopedic and Neurosurgery Spine Surgeons at the Health Sciences Centre in Winnipeg. This encompasses the majority of new and currently managed cases in the Manitoba and Northwestern Ontario.

Subjects will be between the ages of 18 and 90. Male and female subjects will be recruited into the study. All LSS patients will demonstrate intractable neurogenic claudication and radiographically confirmed lumbar spinal stenosis. Exclusion criteria will be any previous lumbar spine surgery, the existence of significant co-morbidity (e.g. neurologic or cardiac condition, disease, etc.) of any form, and any other physical limitations (musculoskeletal injury) preventing the subject from participating in regular activity and the walking program. Subjects participating will be required to speak English.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be between the ages of 18 and 90.
* Male and female subjects will be recruited into the study.
* All LSS patients will demonstrate intractable neurogenic claudication and radiographically confirmed lumbar spinal stenosis.

Exclusion Criteria:

* Any previous lumbar spine surgery, the existence of significant co-morbidity (e.g. neurologic or cardiac condition, disease, etc.) of any form, and any other physical limitations (musculoskeletal injury) preventing the subject from participating in regular activity and the walking program.
* Subjects participating will be required to speak English.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Monitor | 1 week x 4

CONTACTS AND LOCATIONS:
Overall Officials: Michael Johnson, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada